CLINICAL TRIAL: NCT00663949
Title: Phase 2 Trial of Effect of Combine Pentoxifylline and Captopril on Proteinuria in Diabetic Nephropathy
Brief Title: Assessment of the Effect of Captopril Versus Combination of Captopril and Pentoxifylline on Reducing Proteinuria in Type 2 Diabetic Nephropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: shiraz university of medical sciences vice chancellor for research, SUMS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3079
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-03

CONDITIONS: Diabetic Nephropathy
Keywords: diabetes; proteinuria; pentoxifylline
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Proteinuria | interventions — Captopril; Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A,1,II (Active Comparator): patients in this arm takes 25 mg captopril q8h
  Interventions: Drug: Captopril
- A,2,II (Active Comparator)
  Interventions: Drug: Captopril + Pentoxifylline

INTERVENTIONS:
Drug: Captopril — 25 mg captopril tablet q8h
  Arms: A,1,II
Drug: Captopril + Pentoxifylline — patients takes captopril tablets 25 mg q8h and pentoxifylline 400 mg q8h
  Arms: A,2,II

SUMMARY:
Diabetic nephropathy is the most common cause of ESRD and has a great impact on mortality and morbidity of diabetic patients. Despite renoprotective effect of ACE inhibitors in diabetic patients they can not hinder the progression of renal disease completely. Pentoxifylline as a TNFa blocker may hinder progression of diabetic nephropathy in combination of captopril.

DETAILED DESCRIPTION:
Diabetic nephropathy is the most common cause of ESRD and has a great impact on mortality and morbidity of diabetic patients. Despite renoprotective effect of ACE inhibitors in diabetic patients they can not hinder the progression of renal disease completely. TNFa is a cytokine that is a target for medical therapy in diabetic nephropathy. In this study the effect of captopril on overt diabetic nephropathy compared to effect of combination of captopril and an antiTNFa drug ( pentoxifylline).

ELIGIBILITY:
Inclusion Criteria:

1. Absence of kidney or urinary tract disease
2. Absence of high blood pressure OR Controlled blood pressure (≤140/90) with medication other than ACE inhibitors and/or non dihydropyridine calcium channel blockers
3. A well controlled blood sugar level (HbA1c≤7.5%)
4. Adhering to the diet protocol for patients with renal disease

Exclusion Criteria:

1. NYHA functional class III, IV
2. Valvular heart disease
3. Unstable angina, myocardial infarction, cerebrovascular accidents
4. Psychiatric disease
5. Prior allograft kidney transplant
6. Acute illness
7. Infectious disease including urinary tract infection
8. Leukocytosis or any febrile illness at enrollment
9. Prior history or development of any form of malignancy
10. History of alcohol or drug abuse or smoking
11. Pregnancy
12. Need for surgery during the study
13. Allergy to derivatives of methyl xanthines
14. Current Pentoxyphilline use

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
decreasing urinary protein | 2 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Roozbeh, MD, Study Chair — sums; mohammad ghezloo, MD, Study Director — SUMS; mohammad mahdi sagheb, MD, Principal Investigator — SUMS; Amin Banihashemi, Principal Investigator — SUMS
Locations (1):
- Shiraz University of Medical Sciences ,Nemazee and Faghihi Hospital, Shiraz, Fars, Iran